CLINICAL TRIAL: NCT04739423
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind, Crossover, Study of the Pharmacodynamic Effects of CST-103 Co-administered With CST-107 on the Central Nervous System in Subjects With Neurodegenerative Disorders
Brief Title: A Study of Clenbuterol (CST-103) Co-administered With Nadolol (CST-107) in Subjects With Neurodegenerative Disorders
Acronym: CLIN-011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CuraSen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CST103/CST107-CLIN-011
Record Dates: First submitted 2021-01-29; First posted 2021-02-04 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment, Lewy Body Dementia, Parkinson's Disease Rapid Eye Movement Sleep Behavior Disorder, Parkinson's Disease Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Lewy Body Disease | interventions — Clenbuterol; Nadolol

STUDY DESIGN:
Intervention Model Description: Two 14-day periods, 2-way crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CST-103/CST-107 to Placebo (Experimental): Subjects will receive daily doses of CST-103 co-administered with CST-107 for 14 days, followed by a washout period of no drug for 14 days, followed by matching placebo for CST-103 and matching placebo for CST-107 for 14 days.
  Interventions: Drug: clenbuterol (CST-103), nadolol (CST-107), matching placebo
- Placebo to CST-103/CST-107 (Experimental): Subjects will receive daily doses of matching placebo for CST-103 co-administered with matching placebo for CST-107 for 14 days, followed by a washout period of no drug for 14 days, followed by daily doses of CST-103 co-administered with CST-107 for 14 days.
  Interventions: Drug: clenbuterol (CST-103), nadolol (CST-107), matching placebo

INTERVENTIONS:
Drug: clenbuterol (CST-103), nadolol (CST-107), matching placebo — clenbuterol (CST-103) and matching placebo orange capsules; nadolol (CST-107) and matching placebo white capsules

SUMMARY:
This is a Phase II, randomized, placebo-controlled, double-blind, crossover study on the CNS and pharmacodynamic effects of clenbuterol (CST-103) co-administered with nadolol (CST-107) in 4 subject populations with Neurodegenerative Disorders.

DETAILED DESCRIPTION:
Approximately 40 subjects with Parkinson's Disease (PD) with REM Sleep Behavior Disorder (RBD) and Depressive Symptoms, Mild Cognitive Impairment (MCI) with Depressive Symptoms, Dementia with Lewy Bodies (DLB) with Cognitive Fluctuations, and Parkinson's Disease Dementia (PDD) with Cognitive Fluctuations were to be enrolled in a 2 period, 2-way crossover design following study eligibility confirmation during the screening period. The number of subjects enrolled in each cohort could change as emerging data are reviewed from this and other studies.

During each treatment period, subjects received daily doses of clenbuterol (CST-103) co-administered with nadolol (CST-107) or matching placebo for 14 days. Each treatment period was separated by a washout period of 14 days (+5-day window).

All subjects completed clinical and pharmacodynamic assessments during each treatment period and PK blood samples were collected prior to, during and after study medication administration.

ELIGIBILITY:
Inclusion Criteria:

Subjects with PD:

* Male or female subjects ≥ 40 and ≤ 80 years of age, at time of informed consent.
* Diagnosed with Parkinson's Disease, as defined by the United Kingdom Parkinson Disease Brain Bank criteria, associated with REM sleep behavior disorder (PD)
* Modified Hoehn & Yahr ≥ stage 1 and ≤ stage 3 during "On" period as documented in the 3 months prior to Screening or completed at Screening.
* Montreal Cognitive Assessment (MoCA) score ≥ 18 and ≤ 28.

Subjects with MCI:

* Male or female subjects ≥ 50 and ≤ 80 years of age, at time of informed consent.
* Meet the criteria for amnestic Mild Cognitive Impairment (MCI) as per the National Institute on Aging-Alzheimer's Association core clinical criteria.
* Montreal Cognitive Assessment (MoCA) score ≥ 18 and ≤ 26.
* No dementia according to the International Classifications of Diseases (ICD)-10 and Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV.
* Memory complaint reported by the subject or his/her partner, family member or caregiver.
* Score of greater than or equal to one standard deviation below age and educational norms in the Digit Symbol Substitution Test (DSST) during Screening.
* Cognitive decline not primarily caused by vascular, traumatic, or medical problems.

Subjects with Dementia with Lewy Bodies (DLB) or Parkinson's Disease Dementia (PDD):

* Male or female subjects ≥ 50 and ≤ 80 years of age, at time of informed consent.
* Diagnosis of dementia associated with Dementia with Lewy Bodies or Parkinson's disease (PDD).
* Documented cognitive fluctuations endorsed on the Dementia Cognitive Fluctuation Scale (DCFS) with a combined score of ≥8 in items 4, 11, 12 and 14.
* Montreal Cognitive Assessment (MoCA) score ≥ 18 and ≤ 26.
* Have informant or caregiver throughout the study who will submit written consent to cooperate with this study, who routinely accompanies and/or stays with subject 12 hours or more a week, assists with treatment compliance, provides assessments and is able to escort the subject on required visits to study institution.
* Modified Hoehn & Yahr ≥ stage 1 and ≤ stage 3 during "On" period as documented in the 3 months prior to Screening or completed at Screening.
* Stable concomitant medical and/or psychiatric illnesses in the judgement of the PI.

For ALL Subjects:

* Unless confirmed to be azoospermic (vasectomized or secondary to medical cause), males must agree to use a male condom from Day 1 throughout the study when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant.
* Females of childbearing potential (i.e., not postmenopausal or surgically sterile) who have a male partner must have a negative serum pregnancy test result and must agree to one of the following from start of Screening through 30 days after the last study medication administration: use a reliable method of birth control, or monogamous relationship with a male partner of confirmed sterility, or practice complete abstinence.
* Females of non-childbearing potential may be enrolled if it is documented that they are postmenopausal.
* Body weight greater or equal to 50 kg and body mass index (BMI) between 18 and 35 kg/m2, inclusive at Screening.
* Stable medical conditions for 3 months prior to Screening visit (e.g., controlled hypertension, dyslipidemia).
* Willing to follow the protocol requirements and comply with protocol restrictions.
* Capable of providing informed consent and complying with study procedures. Subjects who are unable to provide consent may use a Legally Authorized Representative.

Exclusion Criteria:

* Poorly controlled hypertension despite lifestyle modifications and/or pharmacotherapy.
* Pulmonary disease, including asthma if requiring the use of a β2-Adrenergic bronchodilator, or evidence of clinically significant moderate or severe pulmonary symptoms.
* Clinical signs indicating syndromes such as corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, or Babinski sign.
* Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or meeting DSM-IV diagnostic criteria for psychotic disorders.
* Evidence of any significant clinical disorder or laboratory finding (or in the case of potassium levels below normal range) that renders the participant unsuitable for receiving an investigational drug.
* History of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* Any clinically significant illness or disease as determined by medical and surgical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory assessments conducted at Screening.
* Clinically significant abnormalities of ECG, including QTcF > 450 ms, for males and QTcF > 470 ms for females, and/or HR < 50 beats per minute, or evidence of clinically significant bundle branch blocks, as indicated by 12-lead ECG.
* Calculated creatinine clearance of ≤70 mL/min according to the Cockcroft-Gault equation.
* Current use of any prohibited prescription medication (high-dose aspirin, paracetamol or levodopa, β-AR agonists or β-AR blockers, hypnotics or benzodiazepines other than clonazepam, monoamine oxidase inhibitors, opioids ), over-the-counter medication, or herbal supplements/products.
* Prior treatment with any investigational drug ≤90 days prior to dosing (Day 1), or ≤5 half-lives of the drug (whichever is longer), or current enrollment in any other study treatment or disease study, except for observational studies.
* Known or suspected alcohol or substance abuse within the past 12 months and/or positive test for alcohol or drugs of abuse.
* Active suicidal ideation within 3 months prior to study Screening.
* Positive screening test for hepatitis C antibody (HCV Ab) or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] at Screening).
* Positive screening test for human immunodeficiency virus (HIV).
* Current infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Contraindications to wearing the BioStamp digital device sensors, which include but are not limited to implanted pacemakers, defibrillators, or other active implantable devices.
* Known allergies or hypersensitivities to adhesives or hydrogel.
* Other reasons for which the PI considers it is not in the best interest of the participant to undertake the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — CuraSen Therapeutics, Inc.
Locations (7):
- Australia (3):
  - The University of Sydney, Sydney, New South Wales
  - Wesley Medical Research Ltd, Brisbane, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria
- NZBRI, Christchurch, New Zealand
- United Kingdom (3):
  - MAC, Tankersley, Barnsley
  - MAC, Blackpool, Lancashire
  - MAC, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- PD Sequence 1: Subjects with PD enrolled in Cohort A, randomized to receive CST-103/CST-107 then Placebo
- PD Sequence 2: Subjects with PD enrolled in Cohort A, randomized to receive Placebo then CST-103/CST-107
- MCI Sequence 1: Subjects with MCI enrolled in Cohort A, randomised to receive CST-103/CST-107 then Placebo
- MCI Sequence 2: Subjects with MCI enrolled in Cohort A, randomized to receive Placebo then CST-103/CST-107
- PDD or DLB Sequence 1: Subjects with PDD or DLB enrolled in Cohort B, randomized to receive CST-103/CST-107 then Placebo
- PDD or DLB Sequence 2: Subjects with PDD or DLB enrolled in Cohort B, randomized to receive Placebo then CST-103/CST-107
Period: Overall Study
Arm/Group | PD Sequence 1 | PD Sequence 2 | MCI Sequence 1 | MCI Sequence 2 | PDD or DLB Sequence 1 | PDD or DLB Sequence 2
Started | 12 | 13 | 6 | 7 | 1 | 2
Completed | 12 | 12 | 5 | 7 | 0 | 1
Not Completed | 0 | 1 | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in study.
Groups:
- Overall: All subjects enrolled in study.
Arm/Group | Overall
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  White | 40
Region of Enrollment [Number; unit: participants]
  New Zealand | 15
  United Kingdom | 11
  Australia | 5
  Belgium | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Negative Emotional Bias in the Facial Expression Recognition Task (FERT)
Description: Faces with six different basic emotions (happiness, fear, anger, disgust, sadness, surprise) are briefly displayed on a screen and participants are required to indicate the expression of the face via a button-press. Cohort A only.
Time Frame: Days 7 and 14 of each Treatment Period (Two 14-day periods)
Population: Full Analysis Set (FAS) - The FAS included all randomized study subjects who had taken at least one dose of blinded study drug in this crossover study. In accordance with the protocol this outcome measure was only applicable for Cohort A.
  Data are presented by treatment for each patient population analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- PD - Placebo: Subjects with PD enrolled in Cohort A following treatment with placebo.
- PD - Active: Subjects with PD enrolled in Cohort A following treatment with active.
- MCI - Placebo: Subjects with MCI enrolled in Cohort A following treatment with placebo.
- MCI - Active: Subjects with MCI enrolled in Cohort A following treatment with active.
Arm/Group | PD - Placebo | PD - Active | MCI - Placebo | MCI - Active
Number analyzed (Participants) | 23 | 24 | 12 | 12
Percent change
  Accuracy for happiness - Change from baseline to Day 14 | 8.1316 (2.5783) | 13.6138 (2.5462) | 8.0168 (4.9441) | 6.7407 (4.9441)
  Accuracy for sadness - Change from baseline to Day 14 | -6.9002 (1.7950) | -2.1048 (1.7749) | -7.7744 (2.3576) | -5.8789 (2.3576)
  Reaction time for anger - Change from baseline to Day 7: number analyzed (Participants) | 21 | 23 | 12 | 12
  Reaction time for anger - Change from baseline to Day 7 | -150.77 (78.70) | 16.52 (75.97) | -17.51 (158.55) | -25.03 (165.47)
Statistical Analysis 1: Comparison: PD - Placebo vs PD - Active; Between treatment analysis for Accuracy for happiness - change from baseline to Day 14; Test type: Other; p = 0.0479, Mixed Models Analysis; Least Squares Mean = 5.4822, 95% CI 2-sided [0.0575 to 10.9069]
Statistical Analysis 2: Comparison: PD - Placebo vs PD - Active; Between treatment analysis for Accuracy for sadness - Change from baseline to Day 14; Test type: Other; p = 0.0161, Mixed Models Analysis; Least Squares Mean = 4.7954, 95% CI 2-sided [0.9843 to 8.6064]
Statistical Analysis 3: Comparison: PD - Placebo vs PD - Active; Between treatment analysis of Reaction time for anger - change from baseline to Day 7; Test type: Other; p = 0.0237, Mixed Models Analysis; Least Squares Mean = 167.29, 95% CI 2-sided [25.36 to 309.23]
Statistical Analysis 4: Comparison: MCI - Placebo vs MCI - Active; Between treatment analysis for Accuracy for happiness - change from baseline to Day 14; Test type: Other; p = 0.7188, Mixed Models Analysis; Least Squares Mean = -1.2761, 95% CI 2-sided [-9.2424 to 6.6902]
Statistical Analysis 5: Comparison: MCI - Placebo vs MCI - Active; Between treatment analysis for Accuracy for sadness - Change from baseline to Day 14; Test type: Other; p = 0.5478, Mixed Models Analysis; Least Squares Mean = 1.8955, 95% CI 2-sided [-4.9026 to 8.6935]
Statistical Analysis 6: Comparison: MCI - Placebo vs MCI - Active; Between treatment analysis of Reaction time for anger - change from baseline to Day 7; Test type: Other; p = 0.9510, Mixed Models Analysis; Least Squares Mean = -7.52, 95% CI 2-sided [-291.21 to 276.17]

2. Primary Outcome: Change From Baseline in Cognitive Fluctuations
Description: Dementia Cognitive Fluctuation Scale (DCFS). Number of participants with improvement relative to screening. Cohort B only.
Time Frame: Screening, Days 1 and 14 of each Treatment Period (Two 14-day periods)
Population: All participants enrolled in Cohort B.
Measure: Count of Participants; unit: Participants
Groups:
- PDD or DLB Placebo: Subjects with PDD or DLB enrolled in Cohort B following treatment with Placebo
- PDD + DLB - Active: Subjects with PDD or DLB enrolled in Cohort B following treatment with CST-103/CST-107
Arm/Group | PDD or DLB Placebo | PDD + DLB - Active
Number analyzed (Participants) | 3 | 2
Participants
  How great is the difference between the worst and the best period of function on that day? | 2 | 2
  Length of time sleeping during day. | 2 | 1
  How often is patient drowsy and lethargic during the day? | 1 | 1
  Overall, how would you rate the patient's level of consciousness on a usual day? | 2 | 2

3. Secondary Outcome: Change From Baseline in CANTAB Cognitive Assessments
Description: The CANTAB cognitive assessments consists of a series of interrelated computerized tests of memory, attention, and executive function, administered via a touch sensitive screen. This includes the immediate and delayed Verbal Recognition Memory (VRM) recall and recognition tests that measure the ability to encode and subsequently retrieve verbal information.
Time Frame: Days 1, 7, 14 of each Treatment Period (Two 14-day periods)
Population: Full Analysis Set (FAS) - The FAS included all randomized study subjects who had taken at least one dose of blinded study drug.
  Data are presented by treatment for each patient population analyzed.
Measure: Least Squares Mean (Standard Error); unit: Words
Groups:
- PDD or DLB - Placebo: Subjects with PDD or DLB enrolled in Cohort B following treatment with placebo.
- PDD or DLB - Active: Subjects with PDD or DLB enrolled in Cohort B following treatment with active.
Arm/Group | PD - Placebo | PD - Active | MCI - Placebo | MCI - Active | PDD or DLB - Placebo | PDD or DLB - Active
Number analyzed (Participants) | 25 | 25 | 13 | 13 | 3 | 3
Words
  Immediate Word Recall: Number of words - Change from Baseline to Day 1, 4 hours post dose: number analyzed (Participants) | 25 | 23 | 12 | 13 | 3 | 2
  Immediate Word Recall: Number of words - Change from Baseline to Day 1, 4 hours post dose | -0.50 (0.375) | 0.18 (0.385) | 0.89 (0.531) | 0.83 (0.514) | -1.96 (0.474) | -0.12 (0.514)
  Immediate Word Recall: Number of words - Change from Baseline to Day 14, 4 hours post dose: number analyzed (Participants) | 24 | 24 | 12 | 12 | 2 | 2
  Immediate Word Recall: Number of words - Change from Baseline to Day 14, 4 hours post dose | 0.20 (0.380) | 1.32 (0.380) | 1.89 (0.531) | 1.65 (0.530) | -2.79 (0.514) | -1.29 (0.514)
  Delayed Word Recall: number of words - Change from Baseline to Day 1, 4 hours post dose: number analyzed (Participants) | 25 | 23 | 10 | 12 | 3 | 2
  Delayed Word Recall: number of words - Change from Baseline to Day 1, 4 hours post dose | -2.50 (0.556) | -0.78 (0.572) | 0.64 (0.824) | 0.59 (0.770) | -1.44 (0.431) | 0.51 (0.518)
  Delayed Word Recall: number of words - Change from Baseline to Day 7, 4 hours post dose: number analyzed (Participants) | 23 | 24 | 12 | 12 | 2 | 2
  Delayed Word Recall: number of words - Change from Baseline to Day 7, 4 hours post dose | -1.17 (0.572) | 0.13 (0.564) | 0.37 (0.776) | 1.34 (0.775) | 1.01 (0.518) | 0.01 (0.518)
  Delayed Word Recognition: number of words - Change from Baseline to Day 7, 4 hrs post-dose: number analyzed (Participants) | 23 | 24 | 12 | 12 | 2 | 2
  Delayed Word Recognition: number of words - Change from Baseline to Day 7, 4 hrs post-dose | -1.94 (0.474) | -0.24 (0.466) | -0.44 (0.891) | 0.40 (0.889) | -3.67 (1.109) | -6.17 (1.109)
Statistical Analysis 1: Comparison: PD - Placebo vs PD - Active; Between treatment analysis for Immediate Word Recall: number of words - Change from Baseline to Day 1, 4 hours post-dose; Test type: Other; p = 0.0737, Mixed Models Analysis; Least Squares Mean = 0.68, 95% CI 2-sided [-0.066 to 1.432]
Statistical Analysis 2: Comparison: PD - Placebo vs PD - Active; Between treatment analysis for Immediate Word Recall: number of words - Change from Baseline to Day 14, 4 hours post-dose; Test type: Other; p = 0.0033, Mixed Models Analysis; Least Squares Mean = 1.12, 95% CI 2-sided [0.382 to 1.868]
Statistical Analysis 3: Comparison: PD - Placebo vs PD - Active; Between treatment comparison for Delayed Word Recall: number of words - Change from Baseline to Day 1, 4 hours post-dose; Test type: Other; p = 0.0029, Mixed Models Analysis; Least Squares Mean = 1.72, 95% CI 2-sided [0.600 to 2.840]
Statistical Analysis 4: Comparison: PD - Placebo vs PD - Active; Between treatment analysis for Delayed Word Recall: number of words - Change from Baseline to Day 7, 4 hours post-dose; Test type: Other; p = 0.0247, Mixed Models Analysis; Least Squares Mean = 1.29, 95% CI 2-sided [0.168 to 2.418]
Statistical Analysis 5: Comparison: PD - Placebo vs PD - Active; Between treatment analysis for Delayed Word Recognition: number of words - Change from Baseline to Day 7, 4 hours post-dose; Test type: Other; p = 0.0016, Mixed Models Analysis; Least Squares Mean = 1.69, 95% CI 2-sided [0.653 to 2.732]
Statistical Analysis 6: Comparison: MCI - Placebo vs MCI - Active; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.9126, Mixed Models Analysis; Least Squares Mean = -0.06, 95% CI 2-sided [-1.127 to 1.009]
Statistical Analysis 7: Comparison: MCI - Placebo vs MCI - Active; [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.6570, Mixed Models Analysis; Least Squares Mean = -0.24, 95% CI 2-sided [-1.317 to 0.837]
Statistical Analysis 8: Comparison: MCI - Placebo vs MCI - Active; [analysis description as in outcome 3, analysis 3]; Test type: Other; p = 0.9458, Mixed Models Analysis; Least Squares Mean = -0.06, 95% CI 2-sided [-1.787 to 1.669]
Statistical Analysis 9: Comparison: MCI - Placebo vs MCI - Active; Between treatment analysis for Delayed Word Recall: number of words - Change from Baseline to Day 7, 4 hours post-dose; Test type: Other; p = 0.2327, Mixed Models Analysis; Least Squares Mean = 0.97, 95% CI 2-sided [-0.642 to 2.579]
Statistical Analysis 10: Comparison: MCI - Placebo vs MCI - Active; [analysis description as in outcome 3, analysis 5]; Test type: Other; p = 0.4154, Mixed Models Analysis; Least Squares Mean = 0.84, 95% CI 2-sided [-1.208 to 2.879]

4. Secondary Outcome: Digital Wearable Device (BioStamp) - Sleeping Heart Rate
Description: A wireless device that measures physical activity and sleep while at home.
Time Frame: Screening, Days 1-14 of each Treatment Period (Two 14-day periods)
Population: Per protocol, the BioStamp wearable device was used in a substudy that included only the clinical sites based in Australia and New Zealand. There were a total of 18 subjects in this substudy. However, only 9 subjects provided a dataset that could be analyzed for treatment effect (ie. that included baseline data and end of study period data). Data are presented by treatment for each patient population.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Groups:
- PDD + DLB - Active: Subjects with PDD or DLB enrolled in Cohort B following treatment with placebo
- Overall - Placebo: All subjects following treatment with placebo
- Overall - Active: All subjects following treatment with active
Arm/Group | PD - Placebo | PD - Active | MCI - Placebo | MCI - Active | PDD or DLB - Placebo | PDD + DLB - Active | Overall - Placebo | Overall - Active
Number analyzed (Participants) | 7 | 8 | 0 | 0 | 0 | 0 | 9 | 9
beats per minute | -0.39 (0.466) | 4.59 (0.480) |  |  |  |  | -0.39 (0.394) | 4.67 (0.405)
Statistical Analysis 1: Comparison: Overall - Placebo vs Overall - Active; Between treatment analysis (active - placebo) for Sleeping Heart Rate change from baseline across periods; Test type: Other; p < 0.0001, Mixed Models Analysis; Least Squares Mean = 5.06, 95% CI 2-sided [3.956 to 6.160]

5. Secondary Outcome: Digital Wearable Device (BioStamp) - Sleeping Heart Rate Variability (HRV)
Description: A wireless device that measures physical activity and sleep while at home.
Time Frame: Screening, Days 1-14 of each Treatment Period (Two 14-day periods)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | PD - Placebo | PD - Active | MCI - Placebo | MCI - Active | PDD or DLB - Placebo | PDD + DLB - Active | Overall - Placebo | Overall - Active
Number analyzed (Participants) | 7 | 8 | 0 | 0 | 0 | 0 | 9 | 9
ratio | -0.26 (0.325) | 0.74 (0.330) |  |  |  |  | -0.18 (0.324) | 0.82 (0.329)
Statistical Analysis 1: Comparison: Overall - Placebo vs Overall - Active; Between treatment analysis (active - placebo) for sleeping HRV change from baseline across periods; Test type: Other; p = 0.0017, Mixed Models Analysis; Least Squares Mean = 1.00, 95% CI 2-sided [0.432 to 1.565]

6. Secondary Outcome: Digital Wearable Device (BioStamp) - Sleeping Heart Rate Variability (HRV) - Root Mean Square of Successive Differences (RMSSD)
Description: A wireless device that measures physical activity and sleep while at home.
Time Frame: Screening, Days 1-14 of each Treatment Period (Two 14-day periods)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: RMSSD
Arm/Group | PD - Placebo | PD - Active | MCI - Placebo | MCI - Active | PDD or DLB - Placebo | PDD + DLB - Active | Overall - Placebo | Overall - Active
Number analyzed (Participants) | 7 | 8 | 0 | 0 | 0 | 0 | 9 | 9
RMSSD | 2.40 (3.101) | -7.41 (3.184) |  |  |  |  | -1.16 (3.229) | -11.37 (3.292)
Statistical Analysis 1: Comparison: Overall - Placebo vs Overall - Active; Between treatment analysis (active - placebo) for sleeping HRV root mean square of successive differences change from baseline across periods; Test type: Other; p = 0.0049, Mixed Models Analysis; Least Squares Mean = -10.22, 95% CI 2-sided [-16.867 to -3.567]

ADVERSE EVENTS:
Time Frame: From first dose to end of study visit (approximately 8 weeks).
Description: AEs may have been reported by the subject, discovered through Investigator questioning, or detected through physical examination, laboratory test, or other means.
Groups:
- PD - Placebo: Subjects with PD enrolled in Cohort A receiving placebo.
- PD - Active: Subjects with PD enrolled in Cohort A receiving active.
- MCI - Placebo: Subjects with MCI enrolled in Cohort A receiving placebo.
- MCI - Active: Subjects with MCI enrolled in Cohort A receiving active.
- PDD and DLB - Placebo: Subjects with PDD or DLB enrolled in Cohort B receiving placebo.
- PDD and DLB - Active: Subjects with PDD or DLB enrolled in Cohort B receiving active.
Arm/Group | PD - Placebo | PD - Active | MCI - Placebo | MCI - Active | PDD and DLB - Placebo | PDD and DLB - Active
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/12 | 0/13 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/24 | 0/12 | 0/13 | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 16/25 | 20/24 | 4/12 | 7/13 | 2/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD - Placebo (N=25) | PD - Active (N=24) | MCI - Placebo (N=12) | MCI - Active (N=13) | PDD and DLB - Placebo (N=3) | PDD and DLB - Active (N=2)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD - Placebo (N=25) | PD - Active (N=24) | MCI - Placebo (N=12) | MCI - Active (N=13) | PDD and DLB - Placebo (N=3) | PDD and DLB - Active (N=2)
Headache (Nervous system disorders) | 3 | 5 | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 6 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Parkinsonian rest tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertebral artery anuerysm (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hallucination olfactory (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supine hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Eye oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT04739423/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04739423/SAP_001.pdf